CLINICAL TRIAL: NCT03722173
Title: Relative Bioavailability of a Single Oral Dose of BI 894416 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects (an Open-label, One-way Crossover Study)
Brief Title: A Study in Healthy Men to Test How Itraconazole Influences the Amount of BI 894416 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1371-0004; 2018-002728-17 (EudraCT Number)
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: Open-label, one-way crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 894416 alone (R) / BI 894416+Itraconazole (T) (Experimental): Participants were administered 3 milligram (mg) BI 894416 tablet (1 mg X 3 tablets) orally on Day 1 alone in treatment period 1 (R), and along with 20 milliliter (mL) of 10 mg/ mL Itraconazole oral solution in treatment period 2 (T).
  In period 2 (T), participants received 200 mg ((20 milliliter (mL)) of Itraconazole oral solution once daily for 5 days, from Day -3 to Day 2. On Day 1 participants received additionally after the Itraconazole dosing, 3 mg BI 894416 tablet (1 mg X 3 tablets) orally in treatment period 2 (T). Both treatment periods were separated by a washout period of at least 6 days between BI 894416 administrations. In both treatments, BI 894416 was administered to subjects in the fasting state.
  Interventions: Drug: Itraconazole; Drug: BI 894416

INTERVENTIONS:
Drug: Itraconazole — Oral solution
Drug: BI 894416 — Tablet

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of BI 894416 in plasma when given as oral single dose together with multiple oral doses of itraconazole (Test,T) as compared to when given alone as oral single dose (Reference, R).

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG) and including the neurological examination) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (unless the subject quit smoking for at least 1 year prior to first planned administration of trial medication)
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* History of relevant neurological disorder affecting the peripheral or central nervous system (this includes, but is not limited to: stroke, epilepsy, inflammatory or atrophic diseases affecting the nervous system, cluster headache or any cancer of the nervous system). Febrile seizures in childhood or adolescence, recovered carpal tunnel syndrome, recovered uncomplicated meningitis, recovered herpes zoster, tension headache, occasional benign tics (e.g. due to stress) or minor par- or dysesthesia (e.g. as a side effect of prior blood withdrawal) do not constitute a history of relevant neurological disorder.
* History of immunological disease except allergy not relevant to the trial (such as mild hay fever or dust mite allergy) and except asthma in childhood or adolescence
* History of cancer (other than successfully treated basal cell carcinoma)
* Within 10 days prior to administration of trial medication, use of any drug that could reasonably inhibit platelet aggregation or coagulation (e.g., acetylsalicylic acid)
* Liver enzyme (ALT, AST, gGT) values above upper limit of normal at the screening examination
* History of drug-induced liver injury
* History of heart failure, or any evidence of ventricular dysfunction in the history
* History of hereditary fructose intolerance
* Male subjects with woman of child bearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of first administration of trial medication until 30 days after the last administration of trial medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, two-treatment periods one-way crossover trial in healthy male participants to compare BI 894416+Itraconazole (Treatment(T)) versus BI 894416 alone (Reference(R)). All participants underwent treatment R in Period 1 (Visit 2) and treatment T in Period 2 (Visit 3). There was at least 6 days washout between the administrations of BI 894416.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist site which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Period: Period 1 (2 Days)
Arm/Group | BI 894416 Alone (R) / BI 894416+Itraconazole (T)
Started (Started are treated) | 14
Completed | 14
Not Completed | 0
Period: Washout Period
Arm/Group | BI 894416 Alone (R) / BI 894416+Itraconazole (T)
Started | 14
Completed | 14
Not Completed | 0
Period: Period 2 (4 Days)
Arm/Group | BI 894416 Alone (R) / BI 894416+Itraconazole (T)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who received at least 1 dose of trial medication.
Arm/Group | BI 894416 Alone (R) / BI 894416+Itraconazole (T)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 to the last quantifiable data point is presented. Standard Error (SE) is actually a geometric (g) SE. Pharmacokinetic (PK) samples were collected 3 hours (h) prior dosing and 15 minutes (min), 30 min, 45min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h and 34h after BI 894416 on day 1 of both periods and additionally on 48h and 72h after BI 894416 administration in period 2.
Time Frame: Up to 34 h (period 1) and up to 72 h (period 2) (please refer timeframe in detail in description)
Population: Pharmacokinetic (PK) parameter set (PKS): PKS included all subjects in the TS who provided at least 1 PK parameter that was not excluded because of important protocol deviation (IPDs) relevant to the statistical evaluation the PK endpoints.
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour / Litre (nmol*h/ L)
Groups:
- BI 894416 Alone (R): Participants were administered 3 milligram (mg) BI 894416 tablet (1 mg X 3 tablets) orally on Day 1 alone in treatment period 1 (R).
- BI 894416 + Itraconazole (T): Participants received 200 mg ((20 milliliter (mL)) of Itraconazole oral solution once daily for 5 days, from Day -3 to Day 2. On Day 1 participants received additionally after the Itraconazole dosing, 3 mg BI 894416 tablet (1 mg X 3 tablets) orally.
Arm/Group | BI 894416 Alone (R) | BI 894416 + Itraconazole (T)
Number analyzed (Participants) | 14 | 14
Nanomole*hour / Litre (nmol*h/ L) | 371.77 (1.13) | 526.50 (1.13)
Statistical Analysis 1: Comparison: BI 894416 Alone (R) vs BI 894416 + Itraconazole (T); Point estimates for the ratios of the geometric means (gMeans) (T/R) for AUC0-tz and their 2-sided 90% confidence intervals (CIs) were provided. The difference between the expected means for log(T) - log(R) were estimated by the difference in the corresponding adjusted means (Least Squares Means); Test type: Other — Since the main focus was on estimation and not testing, a formal hypothesis test and associated acceptance range was not specified; no hypothesis was tested; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects for 'subjects' and 'treatment' was used; gMeans ratio (T/R) % = 141.62, 90% CI 2-sided [129.64 to 154.71], Standard Error of Mean 13.30 — Standard error of the mean is actually an intra-individual coefficient variation (CV). Confidence intervals (CIs) were calculated based on the residual error from the ANOVA and quantiles from the t distribution

2. Primary Outcome: Maximum Measured Concentration of BI 894416 in Plasma (Cmax)
Description: Cmax, maximum measured concentration of BI 894416 in plasma is presented. Standard error (SE) is actually geometric (g) SE. Pharmacokinetic (PK) samples were collected 3 hours (h) prior dosing and 15minutes (min), 30 min, 45min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h and 34h after BI 894416 on day 1 of both periods and additionally on 48h and 72h after BI 894416 administration in period 2.
Time Frame: Up to 34 h (period 1) and up to 72 h (period 2) (please refer timeframe in detail in description)
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: Nanomole/ Litre (nmol/ L)
Arm/Group | BI 894416 Alone (R) | BI 894416 + Itraconazole (T)
Number analyzed (Participants) | 14 | 14
Nanomole/ Litre (nmol/ L) | 59.93 (1.07) | 67.91 (1.07)
Statistical Analysis 1: Comparison: BI 894416 Alone (R) vs BI 894416 + Itraconazole (T); Point estimates for the ratios of the gMeans (T/R) for Cmax and their 2-sided 90% CIs were provided. The difference between the expected means for log(T) - log(R) were estimated by the difference in the corresponding adjusted means (Least Squares Means); Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects for 'subjects' and 'treatment' was used; gMeans ratio (T/R) % = 113.32, 90% CI 2-sided [102.47 to 125.32], Standard Error of Mean 15.10 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 894416 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve of BI 894416 in plasma over the time interval from 0 extrapolated to infinity is presented. Standard error (SE) is actually geometric (g) SE. Pharmacokinetic (PK) samples were collected 3 hours (h) prior dosing and 15minutes (min), 30 min, 45min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h and 34h after BI 894416 on day 1 of both periods and additionally on 48h and 72h after BI 894416 administration in period 2.
Time Frame: Up to 34 h (period 1) and up to 72 h (period 2) (please refer timeframe in detail in description)
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: Nanomole*hour / Litre (nmol*h/ L)
Arm/Group | BI 894416 Alone (R) | BI 894416 + Itraconazole (T)
Number analyzed (Participants) | 14 | 14
Nanomole*hour / Litre (nmol*h/ L) | 384.01 (1.13) | 547.36 (1.13)
Statistical Analysis 1: Comparison: BI 894416 Alone (R) vs BI 894416 + Itraconazole (T); Point estimates for the ratios of the gMeans (T/R) for AUC0-∞ and their 2-sided 90% CIs were provided. The difference between the expected means for log(T) - log(R) were estimated by the difference in the corresponding adjusted means (Least Squares Means); Test type: Other — [test comment as in outcome 1, analysis 1]; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects for 'subjects' and 'treatment' was used; gMeans ratio (T/R) % = 142.54, 90% CI 2-sided [130.30 to 155.93], Standard Error of Mean 13.50 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until the individual subject's end of trial date (at least 6 days for period 1 and between 7 and 14 days for period 2).
Description: Treated set (TS): This subject set included all subjects who received at least one dose of study drug.
Groups:
- Itraconazole Alone: Participants were administered 10 mg/ mL Itraconazole oral solution in treatment period 2 only (T). Itraconazole was administered once daily from Day -3 to Day 1 before administration of BI 894416 on Day 1.
Arm/Group | BI 894416 Alone (R) | Itraconazole Alone | BI 894416 + Itraconazole (T)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 8/14 | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 894416 Alone (R) (N=14) | Itraconazole Alone (N=14) | BI 894416 + Itraconazole (T) (N=14)
Diarrhoea (Gastrointestinal disorders) | 0 | 7 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT03722173/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03722173/SAP_001.pdf